CLINICAL TRIAL: NCT06653738
Title: Randomized Placebo-controlled Trial to Assess Efficacies of EMPAgliflozin and Personalized Dietary Counselling for Kidney STONE Prevention in Patients With Calcium Kidney Stones Acronym: EMPASTONE Trial
Brief Title: Trial to Assess the Efficacy of EMPAgliflozin and Personalized Dietary Counseling for Kidney STONE Prevention
Acronym: EMPASTONE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EMPASTONE Trial
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Kidney Stone; Nephrolithiasis; Dietary Exposure
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to either empagliflozin 25 or placebo once daily, and to either personalized or generic dietary counseling (2x2 factorial design).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Empagliflozin and personalized dietary counseling (Experimental): Empagliflozin 25 mg once daily per os and personalized dietary counseling for 3 years
  Interventions: Drug: Empagliflozin 25 MG; Behavioral: Personalized dietary counseling
- Placebo and personalized dietary counseling (Placebo Comparator): Placebo once daily per os and personalized dietary counseling for 3 years
  Interventions: Drug: Placebo; Behavioral: Personalized dietary counseling
- Empagliflozin and generic dietary counseling (Experimental): Empagliflozin 25 mg once daily per os and generic dietary counseling for 3 years
  Interventions: Drug: Empagliflozin 25 MG; Behavioral: Generic dietary counseling
- Placebo and generic dietary counseling (Placebo Comparator): Placebo once daily per os and generic dietary counseling for 3 years
  Interventions: Drug: Placebo; Behavioral: Generic dietary counseling

INTERVENTIONS:
Drug: Empagliflozin 25 MG — Once daily per os for 3 years
  Arms: Empagliflozin and generic dietary counseling; Empagliflozin and personalized dietary counseling
Drug: Placebo — Once daily per os for 3 years
  Arms: Placebo and generic dietary counseling; Placebo and personalized dietary counseling
Behavioral: Personalized dietary counseling — Personalized dietary counseling based on repeat 24-hr urine collections and dietary assessments for 3 years
  Arms: Empagliflozin and personalized dietary counseling; Placebo and personalized dietary counseling
Behavioral: Generic dietary counseling — Generic dietary counseling based on current guidelines without 24-hr urine collection results and without specific dietary assessments for 3 years
  Arms: Empagliflozin and generic dietary counseling; Placebo and generic dietary counseling

SUMMARY:
The aim of this randomized trial with a 2-by-2 factorial design is to test the efficacy of the SGLT2 inhibitor empagliflozin and personalized dietary counseling based on 24-hr urine collection results and dietary assessments for kidney stone recurrence prevention in patients with calcium kidney stones.

Study interventions:

* Empagliflozin 25 mg once daily per os for 36 months
* Personalized dietary counseling for 36 months.

Control interventions:

* Placebo once daily per os for 36 months
* Generic dietary counseling for 36 months.

DETAILED DESCRIPTION:
Background:

Nephrolithiasis is a highly prevalent kidney disorder that causes substantial morbidity, reduced quality of life and enormous healthcare expenditures worldwide. Kidney stones recur frequently, with 10-year recurrence rates of up to 80 %. Existing pharmacological strategies for the prevention of kidney stone recurrence are limited, and dietary counselling practices for patients with kidney stones vary widely. In observational studies and post-hoc analyses of cardiovascular outcome trials, sodium-glucose cotransporter 2 inhibitor (SGLT2i) use was associated with a reduction in kidney stone events in patients with type 2 diabetes. In the recent randomized phase 2 trial SWEETSTONE (NCT04911660), the SGLT2i empagliflozin significantly improved the urinary lithogenic risk profile compared to placebo in non-diabetic patients with calcium kidney stones, by far the most common kidney stone type.

Rationale:

The efficacy of SGLT2is in the prevention of kidney stone recurrence in patients with kidney stones is unknown. Furthermore, the optimal dietary counseling approach for individuals with kidney stones remains unclear.

Objective:

The investigators plan to conduct a 3-year multicentric, double-blind, placebo-controlled factorial trial to assess the efficacy of empagliflozin with either a personalized or generic dietary counselling strategy for recurrence prevention in patients with calcium kidney stones.

Methodology:

The investigators will include 380 adult (≥ 18 years) patients with recurrent (≥ 2 kidney stone episodes in the last 10 years) calcium kidney stones (containing 50% or more of calcium oxalate, calcium phosphate or a mixture of both). Patients with known secondary causes of kidney stones will be excluded. In this randomized trial with a 2-by-2 factorial design, patients will be allocated to either empagliflozin 25 mg or placebo once daily, and to either personalized or generic dietary counselling according to 24-hr urine results. Randomization will be stratified according to the number of kidney stone episodes during the 10 years before enrolment.

The primary endpoint will be radiologic kidney stone recurrence (a composite of stone growth or new stones formed assessed by computed tomography) at 3 years. Secondary endpoints will be symptomatic kidney stone recurrence up to 3 years, and the number of symptomatic recurrences over 3 years. Exploratory endpoints will be changes in blood and urine parameters, vital signs and weight; asymptomatic kidney stone passage; patient-reported pain and quality of life; and kidney stone event-related health care utilization and cost. Safety endpoints assessed will be the frequency of serious adverse events and of pre-defined adverse events of special interest.

ELIGIBILITY:
Inclusion criteria:

1. Written, informed consent.
2. Age 18 years or older.
3. Recurrent kidney stone disease (2 or more stone episodes in the last 10 years).
4. Last kidney stone containing 50% or more of CaOx, CaP or a mixture of both.
5. If taking guideline-recommended medications for kidney stone prophylaxis (e.g. citrate salts) patients must have been on a stable regimen for at least 60 days before randomization, and willing to remain on this stable regimen for the duration of the study.

Exclusion criteria:

1. Patients with a known history of secondary or Mendelian causes of calcium nephrolithiasis
2. Type I diabetes mellitus
3. History of ketoacidosis
4. Treatment with SGLT2 Inhibitor
5. CKD (defined as CKD-EPI eGFR <30 mL/min)
6. Kidney transplant recipient
7. History of recurrent urinary tract infections (>3 episodes/year)
8. Active cancer treatment
9. Less than 3-year life expectancy
10. Pregnancy and breastfeeding
11. Inability to understand and follow the study protocol
12. Known allergy to the study drug
13. Concomitant participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with radiologic stone recurrence | After 3 years
  Radiological stone recurrence is defined as a new stone formed or enlargement of a preexisting stone (assessed by low-dose CT of the kidney at the end of the study compared to the low-dose CT of the kidney at the baseline visit).

SECONDARY OUTCOMES:
Time to symptomatic kidney stone recurrence up to 3 years (time-to-event) | From enrollment to the end of treatment at 3 years
  Symptomatic recurrence is defined as the visible passage of a stone with or without accompanying typical symptoms (such as flank or loin pain and hematuria) or as the presence of a symptomatic or asymptomatic stone that was determined to require surgical removal.
Number of symptomatic stone recurrences per patient (cumulative) | From enrollment to the end of treatment at 3 years
  Symptomatic recurrence is defined as the visible passage of a stone with or without accompanying typical symptoms (such as flank or loin pain and hematuria) or as the presence of a symptomatic or asymptomatic stone that was determined to require surgical removal.

OTHER OUTCOMES:
Changes in blood parameters | From enrollment to the end of treatment at 3 years
  Blood parameters will be measured at screening, Month 3, Year 1, Year 2 and Year 3.
Changes in urine parameters | From enrollment to the end of treatment at 3 years
  24-hr urine analyses will be done at screening, Month 3, Year 1, Year 2 and Year 3.
  Note: results of 24-hr urine analyses will be blinded until the end of the study in patients randomized to generic dietary counselling.
Changes in blood pressure | From enrollment to the end of treatment at 3 years
  Blood pressure measurements will be done at screening, Month 3, Year 1, Year 2 and Year 3.
Changes in weight | From enrollment to the end of treatment at 3 years
  Weight will be measured at screening, Month 3, Year 1, Year 2 and Year 3.
Patient-reported kidney stone-related quality of life | From enrollment to the end of treatment at 3 years
  Patient-reported kidney stone-related quality of life will be assessed by the Wisconsin Stone-Quality of Life (WSQoL) questionnaire at baseline, Month 3, Year 1, Year 2 and Year 3. Higher scores indicate better quality of life.
Patient-reported health-related quality of life (HRQoL) | From enrollment to the end of treatment at 3 years
  Patient-reported HRQoL will be assessed by using the short form-36 version 2 (SF-36v2) questionnaire at baseline, Month 3, Year 1, Year 2 and Year 3. Higher scores indicate higher HRQoL.
Number of patients with asymptomatic kidney stone passage | At 3 years
  Asymptomatic passage is defined as a stone present on the baseline CT but not on the end of study CT without causing any symptoms in the patient.
Kidney stone-related health care utilization | From enrollment to the end of treatment at 3 years
  Data on emergency visits, hospitalizations and doctoral visits in relation to kidney stone disease
Kidney stone-related cost | From enrollment to the end of treatment at 3 years
  Total kidney stone-related cost (direct and indirect).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fuster, Principal Investigator — Inselspital, Bern University Hospital
Locations (21):
- France (2):
  - University Hospital Amiens-Picardie, Amiens
  - Hôpital Tenon, Paris
- Charité University Medicine Berlin, Berlin, Germany
- Verona University Hospital, Verona, Italy
- Switzerland (17):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - University Hospital Basel, Basel
  - Regionalspital Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Chur, Chur
  - Kantonsspital Fribourg, Fribourg
  - University Hospital Geneva (HUG), Geneva
  - Lausanne University Hospital (CHUV), Lausanne
  - Kantonsspital Luzern, Lucerne
  - Regionalspital Lugano, Lugano
  - Kantonsspital Neuchâtel, Neuchâtel
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Sion, Sion
  - Kantonsspital Solothurn, Solothurn
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No
Once results have been published, trial data will be accessible to external researchers and coded datasets corresponding to each publication will be made available. Investigators wishing to replicate the analyses or to do an individual patient meta-analysis may request the data to the Sponsor-Investigator.

REFERENCES:
- [Background] Schietzel S, Bally L, Cereghetti G, Faller N, Moor MB, Vogt B, Rintelen F, Trelle S, Fuster D. Impact of the SGLT2 inhibitor empagliflozin on urinary supersaturations in kidney stone formers (SWEETSTONE trial): protocol for a randomised, double-blind, placebo-controlled cross-over trial. BMJ Open. 2022 Mar 14;12(3):e059073. doi: 10.1136/bmjopen-2021-059073. PMID 35288397